CLINICAL TRIAL: NCT06785402
Title: Phase 1/2, Randomized, Double-Blind, Placebo-Controlled Trial of Pulse Dosed Ceftriaxone for Post-Treatment Lyme Disease
Brief Title: Ceftriaxone for Post-Treatment Lyme Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Columbia Clinical Trials Network for Lyme and Other Tick-Borne Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2024-0373
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Post-Treatment Lyme Disease Syndrome
Keywords: Post-Treatment Lyme disease Syndrome (PTLDS); Ceftriaxone; Persistent Symptoms
MeSH Terms: conditions — Post-Lyme Disease Syndrome

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized 1:1 receiving either pulse-dosed ceftriaxone or placebo [dextrose (5% in water), (D5W)], intravenously. Subjects will be follow-up phase out to 12 months. Subjects will be unblinded at 6 months and those randomized to the placebo group will be offered pulse-dosed ceftriaxone on the same schedule as those randomized to the drug group. All subjects will be followed up for a total of 12 months post treatment initiation.
Who Masked: Participant, Investigator
Masking Description: Participants and the study team will be blinded. The research pharmacist will be the unblinded party.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceftriaxone 2 GM (Experimental): Administration of IV ceftriaxone or D5W. Subjects will be infused approximately every 5 days (+/- 1 day) over the course of ~6 weeks. Subjects will receive a total of 9 infusions throughout the treatment phase of the study, with the last infusion tentatively scheduled for Day 41 (+/- 3 days).
  Interventions: Drug: Ceftriaxone treatment
- Placebo (Placebo Comparator): Placebo [dextrose (5% in water), (D5W)] IV following the same infusion schedule as the ceftriaxone arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ceftriaxone treatment — 9 infusions spaced out approximately every 5 days
  Arms: Ceftriaxone 2 GM
Drug: Placebo — D5W (placebo)
  Arms: Placebo

SUMMARY:
Lyme disease is a public health crisis in the US. It is estimated that over 400,000 cases occur every year with 10-20% of those infected going on to develop Post-Treatment Lyme disease Syndrome (PTLDS). The goal of this study is to investigate if giving Ceftriaxone every 5 days for about 6 weeks kills the organism that produces persistent Lyme infection.

Enrolled participants will be randomized 1:1 receiving either pulse-dosed ceftriaxone or placebo [dextrose (5% in water), (D5W)], intravenously. Participants will be evaluated at each of the study visits, and then in a follow-up phase out to 12 months. They will be unblinded at 6 months and those randomized to the placebo group will be offered pulse-dosed ceftriaxone on the same schedule as those randomized to the drug group. All patients will be followed up for a total of 12 months post treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years at the time of consent
* Ability and willingness to sign informed consent
* Available for the study period
* Must have met the definition of a prior well-defined or probable Lyme disease infection, AND meet the definition of PTLDS
* Provide consent for release of medical history records and photographs from primary care physician, college or university, urgent care or emergency room visit
* Have a level of fatigue that interferes with their ability to function in their job, schooling, or other social/personal activities (FSS score of 4 or higher)
* Subjects will need to have been off of antibiotics (those standard antibiotics used to target Lyme disease to include doxycycline, amoxicillin, cefuroxime, azithromycin, ceftriaxone or penicillin) for at least 6 weeks prior to study enrollment and be willing to remain off of any outside antibiotics during the duration of the treatment component of the study.

Exclusion Criteria:

* Female: pregnant or lactating
* Women who intend to become pregnant during the treatment study period (approximately 45 days)
* Patients with a diagnosis of Lyme disease based on only a positive Lyme IgM immunoblot
* A history of cephalosporin allergy or significant intolerance
* Lyme related symptoms that have been present for greater than 10 years
* Blood tests confirming infection with human immunodeficiency virus- 1 (HIV-1), hepatitis C, hepatitis B (assessed by HbsAg) virus.

Note: Subjects who have well controlled HIV, who are on ART with a CD4 count of >200 will be allowed to participate.

* Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition to include any finding of increased suicide risk per the CSSRS scale (score 6 or greater), which in the opinion of the investigator prevents the subject from participating in the study
* Known concurrent rheumatologic or similar disease thought to interfere with study participation or confound results at the discretion of the investigator. These may include but are not limited to rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, psoriasis, fibromyalgia, chronic fatigue syndrome/myalgic encephalomyelitis, or obstructive sleep apnea
* Hives, shortness of breath, swelling of the lips or throat, or hospitalization related to a previous treatment with a cephalosporin antibiotic, or severe allergic reaction to penicillins (e.g. anaphylaxis or severe rash with Stevens Johnson syndrome or similar)
* Planned travel during the study period that would interfere with the ability to complete all study visits (this can be a temporary exclusion with plan to schedule enrollment during a window of time during which they could attend their study visits)
* Significant screening physical examination abnormalities or chronic medical condition that in the opinion of the investigator may impact subject safety
* Participation (active or follow-up phase) or planned participation in another vaccine, drug, or medical device in the 4 weeks prior to this trial or during the trial
* Prior history of Clostridium difficile infection
* Unable to comply with study requirements
* Clinician discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of pulse-dosed ceftriaxone | 12 months post treatment initiation
  To assess the safety of pulse-dosed ceftriaxone in PTLDS when compared to placebo as well as historical data based on the number of reported adverse and serious adverse events.
Tolerability of pulse-dosed ceftriaxone | 12 months post treatment initiation
  To assess the tolerability of pulse-dosed ceftriaxone in PTLDS when compared to placebo as well as historical data based on the number of reported adverse and serious adverse events.
Study Feasibility | 6 month enrollment period
  To assess the recruit the patients within the pre-determined period of time (6 months).

SECONDARY OUTCOMES:
Clinical Improvement - Physical and mental summary indices | 12 months post treatment initiation
  To assess clinical improvement after treatment using additional clinical outcome measures. Primary functional change with the physical and mental summary indices of the SF-36 as either responder or non-responder (a change of 6.5 points on the SF-physical health summary scale, and 7.9 points on the mental health summary scale respectively). Eight scales are used and when combined measure the physical and mental health of participants. Each scale is scored to have same average (50) and the same standard deviation (10 points). with a score below 50 representing below average health.
Clinical Improvement - General Symptom Questionnaire (GSQ-30) | 12 months post treatment initiation
  To assess clinical improvement after treatment using additional clinical outcome measures. General Symptom Questionnaire (GSQ-30).GSQ-30 us used to assess symptom burden and specifically pain/fatigue, neuropsychiatric, neurologic, and viral-like symptom burden impacting function. Each symptom is measured on scale of 0 (not at all) to 4 (very much) for an overall score of 0-120 with higher scores representing higher burden.
Clinical Improvement - PROMIS-29 | 12 months post treatment initiation
  To assess clinical improvement after treatment using additional clinical outcome measures using PROMIS-29 which has multiple sections and scoring varies by section.
  The min/max are as follows: Physical Function (PF) 4-20, Anxiety 4-20, Depression 4-20, Fatigue 4-20, Sleep Disturbance- 4-20, Ability to Participate in Social Roles and Activities (APSRA) 4-20, Pain Interference 4-20, Pain Intensity 0-10.
  For PF and APSRA, improvement would be tracked by an increase in score. For Anxiety, Depression, Fatigue, Sleep Disturbance, Pain interference, and Pain Intensity improvement would be tracked by a decrease in score.
  A higher score in PF and APSRA suggest better health. A higher score in Anxiety, Depression, Fatigue, Sleep Disturbance, Pain interference and Pain Intensity suggests lower health.
  A score change of 5 points or more is considered clinically meaningful.
Clinical Improvement - Quantitative Lyme VlsE1/pepC10 Ab | 12 months post treatment initiation
  To assess clinical improvement after treatment using additional clinical outcome measures changes in quantitative Lyme VlsE1/pepC10 Ab. Higher titers represent higher antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Bindu Balani, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No